CLINICAL TRIAL: NCT00337623
Title: Corticosteroids and Cataracts : Prospective Study of the Impact of Systemic Corticosteroid Therapy on Lens Transparency Evaluated by Scheimpflug Photography and Quantification of Lens Autofluorescence.
Brief Title: Impact of Systemic Corticosteroid Therapy on Lens Transparency and Quantification of Lens Autofluorescence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU63-0011
Record Dates: First submitted 2006-06-01; First posted 2006-06-16 (Estimated); Last update posted 2006-06-23 (Estimated); Status verified 2006-06

CONDITIONS: Patients With Systemic Inflammatory Diseases Receiving for the First Time a Protracted General Corticostroid Therapy
Keywords: Cataracts; Corticosteroids; Scheimpflug; Lens autofluorescence
MeSH Terms: conditions — Cataract | interventions — Prednisolone

INTERVENTIONS:
Drug: Prednisolone

SUMMARY:
Corticosteroid therapy is usually regarded as a risk factor for the development of posterior subcapsular cataracts but prospective studies on this topic and accurate assessment of this potential adverse effect are lacking. We will evaluate changes of lens transparency after administration of systemic corticosteroid therapy for at least one year with Scheimpflug photography and quantification of lens autofluorescence.

DETAILED DESCRIPTION:
Corticosteroid therapy is usually regarded as a risk factor for the development of posterior subcapsular cataracts but prospective studies on this topic and accurate assessment of this potential adverse effect are lacking. We will evaluate changes of lens transparency after administration of systemic corticosteroid therapy for at least one year with Scheimpflug photography and quantification of lens autofluorescence.

ELIGIBILITY:
Inclusion Criteria:

* Patient who starts a treatment with Prednisone, Prednisolone or Methylprednisolone for an Expected time of one year at least, with normal lens autofluorescence at inclusion.

Exclusion Criteria:

* Previous cataracts and abnormal increase of lens autofluorescence considering age
* Previous elevation of intraocular pressure
* Progressive inflammatory or non inflammatory ocular disease
* Eye drop except artificial tears
* Insulin dependent and non insulin dependent diabetes
* Atopic dermatitis
* Previous protracted corticosteroid therapy
* Drugs known to be associated with an increased risk of cataract

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2000-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Cataracts on Ophthalmologist's Examination
Increase of Lens Autofluorescence
Increase of Lens Density on Scheimpflug Photography

SECONDARY OUTCOMES:
Potential risk factor of cataracts related to the underlying disease or the individual
Potential effect of time allowed from the beginning of treatment, duration and dosage of corticosteroids.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Andre, Doctor, Principal Investigator — University Hospital, Clermont-Ferrand; Olivier Aumaitre, Doctor, Principal Investigator — Hopital Gabriel Montpied (Clermont-Ferrand)
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France